CLINICAL TRIAL: NCT07049679
Title: A Lifestyle Change Program for Managing Diabetes Among the Marshallese in Northwest Arkansas: A Pilot Trial
Brief Title: A Lifestyle Change Program for Managing Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial phase of the research program was denied funding.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 298932
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care - Group B (No Intervention): This group will not participate in the AHD Program. The group participants will continue their routine care but will be invited to all 6 sessions on managing a healthy diet run by the EFNEP team.
- ActiveHeal Diabetes (AHD) Program - Group A (Experimental): This group will continue routine care and participate in the AHD Program. AHD Program.
  Interventions: Behavioral: ActiveHeal Diabetes (AHD) Program

INTERVENTIONS:
Behavioral: ActiveHeal Diabetes (AHD) Program — Biweekly phone/Zoom calls to support physical activity and dietary behavior change, focused on history, experience, benefits and adaptation
  Arms: ActiveHeal Diabetes (AHD) Program - Group A

SUMMARY:
The proposed study aims to fill the gap by adapting an evidence-based intervention and conducting a pilot trial to determine the new program's estimated effect sizes on occupational resilience, A1c, and diabetes-related quality of life. Developing and adapting Lifestyle Redesign (LR) for Marshallese diabetes management is significant because it would reduce health disparities in a community that is disproportionately affected by the disease, and a large number of Marshallese (currently approximately 15,000) have resided in the northwest Arkansas region since the 1980s.

DETAILED DESCRIPTION:
To pilot-test AHD Program, a lifestyle change intervention for diabetes management, and obtain estimates of effect sizes on occupational resilience, A1C, and diabetes-related quality of life. It is hypothesized that occupational resilience, diabetes-related quality of life, and A1C will be improved by the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Marshallese Adults
* type 2 diabetes and test results (within 30 days) showing A1C greater than 6.4% or Estimated Average Glucose greater than 137 mg/dL.
* Able (and willing) to participate in exercise, diet management, and group dancing.

Exclusion Criteria:

* Marshallese who otherwise meet inclusion criteria but are not willing to commit to active participation in a lifestyle change intervention.
* Comorbidities that limit participation in the specified activities (i.e., stepper exercises, dieting, and dancing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-06 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Occupational Resilience Measure (ORM 1.0) | At time of enrollment and week 15
  a 20-item self-report assessment designed to evaluate occupational resilience, which is the capacity to persist in an occupation despite adversity
Diabetes-related quality of Life (RV-DQOL) | At time of enrollment and week 15
  The primary objective of the RV-DQoL is to measure various aspects of quality of life affected by diabetes, including:
  Satisfaction: Assessing patient satisfaction with different aspects of their life, including time spent managing diabetes and receiving checkups, current treatment, knowledge about diabetes, body appearance, and overall life satisfaction.
  Impact: Evaluating the extent to which diabetes impacts daily life, including feelings of physical illness or pain related to treatment, embarrassment related to managing diabetes in public, and interference with family life.
  Worry: Assessing the degree of worry related to diabetes, such as passing out due to low blood sugar, changes in body appearance, and the potential for developing complications.
A1C lab measure | screening and week 15
  is a blood test that measures your average blood sugar (glucose) levels over the past two to three months. It works by measuring the amount of glucose attached to hemoglobin, a protein in your red blood cells responsible for carrying oxygen.

IPD SHARING:
Plan to Share IPD: No